CLINICAL TRIAL: NCT02272179
Title: Brief Intervention for Suicide Risk Reduction in High Risk Adolescents
Acronym: ASAP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Brent, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH100451 (NIH)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Adolescent Behavior
Keywords: adolescence; suicidality; depression
MeSH Terms: conditions — Adolescent Behavior; Suicidal Ideation; Depression | interventions — cellu-brite; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ASAP Treatment and Brite (Experimental): Participants in the experimental arm received the ASAP treatment, during their transition from inpatient to outpatient care, as well as the Brite app for distress tolerance/emotion regulation and safety planning.
  Interventions: Behavioral: As Safe As Possible; Behavioral: Brite
- Treatment as Usual (Active Comparator): Participants in this grouping were studied as they proceed from inpatient to outpatient care, per usual treatment protocols at each site. Participants completed paper safety plans as part of their regular treatment, which is a standard of care for suicidal youth.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: As Safe As Possible — The ASAP (As Safe As Possible) treatment is a brief, intensive intervention initiated during inpatient care and transitioning to outpatient care. The intervention focuses on 1) using motivational interviewing (MI) strategies throughout care; 2) developing a safety plan, including adapting the plan to an interactive safety plan phone app, Brite); and 3) using treatment modules to target specific risk factors that are selected based on individual need.
  Other Names: ASAP
  Arms: ASAP Treatment and Brite
Behavioral: Brite — Brite is a HIPAA-compliant mobile application designed to provide the participants with emotion regulation and distress tolerance skills, social support, and convenient access to safety plan resources via the patients' phone.
  Arms: ASAP Treatment and Brite
Behavioral: Treatment as Usual — Participants received usual treatment for suicidal adolescents as they transition from inpatient hospitalization to outpatient therapy, which included a paper safety plan.
  Arms: Treatment as Usual

SUMMARY:
Adolescent suicide is the 2nd leading cause of death in this age group. There are no validated treatments to decrease the risk of adolescent suicidal behavior, and there are especially no interventions to target the highest risk period for adolescent suicide and suicidal behavior, namely during the time of transition from inpatient to outpatient care. This purpose of this project was to develop a novel, brief intervention that can be delivered on an inpatient unit prior to the transition to outpatient care, and augment known factors to protect adolescents from suicidal behavior, and extend the impact of treatment by liaison with the outpatient therapist and the development of a personalized safety plan phone application. This treatment, ASAP, focuses on augmenting adherence to the components of ASAP and outpatient aftercare, development of a personalized Safety Plan, and Affect Protection, through helping the teen and family promote a positive mood, tolerate distress, engage in healthy emotion regulation and access social support.

DETAILED DESCRIPTION:
This 2-site R34 project developed a brief, flexible, manualized intervention with supporting phone app with the purpose of reducing the risk of suicidal behavior in adolescents with high suicidal ideation or a recent suicide attempt, during the transition from inpatient to outpatient care. This transition period is the highest risk period for attempted and completed suicide. Suicide is the 2nd leading cause of adolescent mortality, and there are currently no established interventions for suicidal teens. By developing a treatment that can be delivered on an inpatient unit prior to the transition to outpatient treatment, we anticipated being able to lower suicidal risk and increase the likelihood that participants will attend subsequent outpatient treatment. In keeping with the priorities of NIMH, this intervention aimed at reducing the risk of suicide and suicidal behavior was trans-diagnostic. We term the intervention ASAP, with anticipated components: (1) Adherence-promoting engagement and adherence to treatment through motivational interviewing; (2) Safety planning; and (3) Affect Protection- selecting from a menu of techniques for maintaining positive affect (e.g. savoring and switching strategies, mobilizing social support, engaging in emotion regulation and distress tolerance skills). Each of these components was delivered within a Motivational Interviewing framework for enhancing intrinsic motivation for change. Treatment was brief (3-5 hours), and flexibly delivered on inpatient units prior to initiation of outpatient treatment.

ASAP included the family in the treatment, and a safety plan phone app to extend the impact of treatment was also developed. Innovative features included: (1) delivery of an intervention at a time and place when suicidal risk is highest; (2) augmentation of protective factors against recurrent suicidal behavior, specifically by promoting development of positive affect, emotion regulation, distress tolerance, and social support; (3) a Safety plan phone app to extend the impact of treatment; and (4) liaison with the outpatient therapist to ensure continuity of care.

This project conducted an RCT of ASAP followed by Aftercare (AC) vs. AC alone to determine ASAP's feasibility, acceptability, impact on proximal targets (e.g., adherence to outpatient care, sleep, positive affect, substance use), suicidal ideation and behavior. In total 68 suicidal adolescents were enrolled, 2 of whom were withdrawn following baseline assessment and were excluded from analyses, resulting in the final study sample size of 66. ASAP, developed with and intended for community clinicians, has the potential to be a sustainable intervention to reduce the burden of adolescent suicidality. Data analyses have been completed and results are being finalized.

ELIGIBILITY:
Inclusion Criteria:

* Child participants will be adolescents (aged 12-17.11 years) admitted to an inpatient unit for a recent suicide attempt or significant suicidal ideation with a plan or intent. We define a suicide attempt, as per the Columbia Clinical Algorithm for Suicide Assessment (C-CASA), as "self-destructive behavior with inferred or stated intent to die."
* Participants must be English-speaking.
* Participants can have unipolar or bipolar disorder, conduct or oppositional disorder, eating disorder, or alcohol or substance use or abuse or dependence.

Exclusion Criteria:

* Child participants to be excluded will be those with current psychosis, mania, <90% of ideal body weight, or IQ<70 (based on the age-appropriate Wechsler Intelligence Scale if concerns about intellectual capabilities are evident at assessment), as these conditions may require more intensive interventions or limit comprehension of the intervention components.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Suicidal behavior and ideation | Weeks 4, 12, and 24
  Suicidal attempts were the major outcome and secondarily, suicidal ideation. Information about past and current suicidal behavior was obtained using the Columbia Suicide History Form, with ideation and behavior classified using the Columbia Suicide Severity Rating Scale (CSSRS). Self-reported ideation was assessed using the Suicidal Ideation Questionnaire - Junior (SIQ-Jr). The two main outcomes, assessing recurrent suicidal behavior and change in suicidal ideation, was assessed at weeks 4, 12, and 24.

SECONDARY OUTCOMES:
Course of disorder and AC treatment. | Weeks 4, 12, and 24
  Attendance to treatment and type of treatment was documented by the Treatment History Form. The electronic medical record and Youth Self Report will also be used to document the presence of psychiatric disorders. The Treatment History Form derives forms of treatment demonstrated on the Child and Adolescent Services Assessment (CASA) using the structure of the Adolescent Longitudinal Interval Follow-up (A-LIFE).
Treatment target: motivation for treatment | Weeks 4, 12, and 24
  Participants rated readiness on a 1-10 scale to assess Readiness to change, Importance of change, and Confidence in ability To Change with regard to coping with suicidal urges [RICTC].
Treatment target: positive and negative affect | Weeks 4, 12, and 24
  Positive and negative affect was monitored by the Positive and Negative Affect Scale [PANAS]).
Treatment target: emotion regulation | Weeks 4, 12, and 24
  Emotion regulation was measured by the Regulation of Emotions Questionnaire.
Treatment target: distress tolerance | Weeks 4, 12, and 24
  Distress tolerance was measured by the Distress Tolerance Scale.
Treatment target: social support | Weeks 4, 12, and 24
  Perceived social support was assessed using the Multidimensional Scale of Perceived Social Support (MSPSS).
Client Satisfaction | Weeks 4, 12, and 24
  Client Satisfaction about ASAP was obtained from the patient and a caretaking parent using the Client Satisfaction Questionnaire-8 (CSQ-8), which has been used in other adolescent treatment studies and has high internal consistency (coefficient α = .93). We also adapted the Computer System Usability Scale (CSUQ) to assess satisfaction with the phone app. The CSUQ was completed by the participant, and is based on earlier measures designed to predict the adoption of technology, based on two main factors: ease of use (easy to learn, access, flexibility, quality of sound, quality of visual display) and usefulness (able to access when needed, helpful when used), scored along 7-point Likert Scales.
Qualitative Interviews | Weeks 4, 12, and 24
  With Dr. Lee's guidance, we conducted brief semi-structured exit interviews following the intervention with both the parent and teen, which were developed and coded on the basis of our original qualitative interviews, to assess the acceptability of treatment. In these interviews, we obtained feedback about perceived effectiveness of the components of treatment, the appropriateness of treatment targets, identification of other targets or approaches that would have been more helpful, barriers to participation, and utility of the phone apps. The phone app was designed to track how often the participant used the apps and what components were accessed. We obtained similar feedback from the ASAP clinicians and from the outpatient aftercare therapists. Based on exit interviews, participant satisfaction, and outcome data from the open trial, we modified the manual and app.

CONTACTS AND LOCATIONS:
Overall Officials: David Brent, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwest, Dallas, Texas

REFERENCES:
- [Result] Kennard BD, Biernesser C, Wolfe KL, Foxwell AA, Craddock Lee SJ, Rial KV, Patel S, Cheng C, Goldstein T, McMakin D, Blastos B, Douaihy A, Zelazny J, Brent DA. Developing a Brief Suicide Prevention Intervention and Mobile Phone Application: a Qualitative Report. J Technol Hum Serv. 2015 Oct 1;33(4):345-357. doi: 10.1080/15228835.2015.1106384. Epub 2015 Dec 14. PMID 26977137
- [Result] Kennard BD, Goldstein T, Foxwell AA, McMakin DL, Wolfe K, Biernesser C, Moorehead A, Douaihy A, Zullo L, Wentroble E, Owen V, Zelazny J, Iyengar S, Porta G, Brent D. As Safe as Possible (ASAP): A Brief App-Supported Inpatient Intervention to Prevent Postdischarge Suicidal Behavior in Hospitalized, Suicidal Adolescents. Am J Psychiatry. 2018 Sep 1;175(9):864-872. doi: 10.1176/appi.ajp.2018.17101151. Epub 2018 Jul 19. PMID 30021457
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793